CLINICAL TRIAL: NCT04544709
Title: Intradiscal Platelet-Rich Plasma Injection for Chronic Discogenic Low Back Pain
Brief Title: Intradiscal Platelet Rich Plasma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Zack McCormick, Zachary McCormick, MD FAAPMR, Associate Professor, Director of Clinical Spine Research, Director of Interventional Spine and Musculoskeletal Medicine Fellowship, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 117455
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Discogenic Pain; Low Back Pain; Chronic Pain
Keywords: Platelet Rich Plasma
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Discogenic Low Back Pain (Other): Patient with Refractory Discogenic Low back pain who will be scheduled for platelet rich plasma injection as standard of care.
  Interventions: Drug: Low back intradiscal injection of platelet rich plasma (PRP)

INTERVENTIONS:
Drug: Low back intradiscal injection of platelet rich plasma (PRP) — SOC Intradiscal Lumbar PRP Procedure : A small amount of blood is drawn from you, then it is spun in a centrifuge to obtain only the platelets and few other cells. After being spun the small amount of platelets will be injected into the specific disc that is believed to be causing pain in an attempt to help reduce inflammation and pain at the site. The injection will be done under fluoroscopic guidance (x-ray) that allows very careful and precise placement of the needle.

SUMMARY:
To assess changes in pain and function in patients with discogenic low back pain after a standard of care intradiscal injection of Platelet-Rich Plasma (PRP).

DETAILED DESCRIPTION:
Low back pain is one of a few conditions which affects all individuals through the lifespan. The etiology of low back pain is multifactorial and in many cases self-limiting, however it also is the leading cause for working age adults to be disabled with more than $87 billion spent on low back pain disorders in 2013 Lumbar disc herniation and internal disc disruption are two causes more common in these younger age groups reaching 39-42% with a predicted probability above 60% until age 50y. While the natural history of disc herniation suggests most individuals will return to a prior level of function in 3-6 months, there is a high rate of recurrent episodes which can cause short-term disability. Continued pain from a discogenic source can lead to decreased activity levels and accelerate degenerative changes in the disc and facet joints as described by Kirkaldy-Willis.

Current guidelines for treatment of axial low back pain from discogenic sources including those with radiculopathy include a 6-12-week course of conservative care including medications, therapy, acupuncture, chiropractic and exercise before an interventional paradigm of injections and/or surgical treatment. For those individuals who do not improve with conservative care and have predominately axial pain, options are limited as success rates from epidural steroid injections and surgery are 50% or less. Other treatments include chymopapain injection, intradiscal electrothermal annuloplasty (IDET), nucleoplasty, methylene blue injection, ozone injection , fibrin sealant injections. All of which have 50% or less likelihood of reducing pain more than 50%, although much of this data is from uncontrolled or prospective case-control studies only.

Platelet- rich plasma (PRP) injections stand apart from those listed above in that they are purported to be "regenerative" interventions for the diseased lumbar disc. PRP is a concentrated injectant of growth factors and anabolic factors which have in vitro and animal studies that have demonstrated upregulated proteoglycan synthesis and nucleus pulposus proliferation, restoration of disc height, healing of annular puncture wounds and anti-inflammatory effect with down regulation of TNF-alpha and IL-1. There has been limited clinical trials in humans on the effect of intradiscal PRP, including 3 trials of which 1 is a RCT and 2 are prospective series. Efficacy of intra-discal injection has shown statistically significant benefits in reduction in pain, improvement in physical function at follow-up points from 3-24 months. Each of these trials have limited sample sizes, short duration follow-up and lack of a standardized PRP preparation, making the generalizability difficult.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years of age at day of enrollment.
2. Clinical diagnosis of refractory discogenic low back pain for >3 months.
3. Magnetic resonance imaging pathology consistent with clinical symptoms/signs or positive lumbar provocative discography according to SIS/IASP standards at one or two levels.
4. Back pain greater than leg pain with an intensity of at least 4/10 or higher using the Numerical Rating Scale (NRS).
5. Pain duration of more than 12 weeks despite trial of conservative therapy (medications, physical therapy, or chiropractic care) for 2 months.

Exclusion Criteria:

1. Refusal to participate, provide consent, or provide follow-up information for the 24-month duration of the study.
2. Contraindications to intradiscal injection of PRP (active infection, bleeding disorders, current anticoagulant or antiplatelet medication use, allergy to iodinated contrast, penicillin or clindamycin and pregnancy or breastfeeding).
3. More than 2 levels of clinical or discogram proven pain.
4. Non-discogenic source of low back pain as identified by separate diagnostic blocks.
5. Negative lumbar provocation discography.
6. Active moderate to severe lumbar radiculopathy.
7. Intradural disc herniation.
8. Spinal fracture within the past 6 months.
9. Steroid injection in the spine within the last 30 days.
10. Any intradiscal injection other than contrast dye or anesthetic in the last 30 days.
11. Prior fusion at level considered to be the source of the pain.
12. Prior lumbar spine surgery within the last 6 months.
13. AP diameter of spinal canal less than or equal to 9mm at level to be treated.
14. Severe uncontrolled medical condition.
15. Moderate to severe hepatic dysfunction.
16. Severe psychological illness.
17. History of Inflammatory arthritis.
18. Malignancy within past 5 years except basal cell or squamous cell skin cancer.
19. Current use of equal to greater than 30mg morphine-equivalent per day of opioid use.
20. A history of alcohol or drug abuse within past 5 years.
21. Use of any investigational drug within past 30 days.
22. A known allergy or sensitivity to citrate (used for processing PRP).
23. Severe anaphylactic/anaphylactoid reaction to any medications used.
24. Pending litigation involving subject's back pain.
25. No insurance coverage for any subsequent tests or procedures.
26. Disc protrusion greater than 5mm from base of vertebral body.
27. Greater than 50% disc height loss at involved level(s).
28. Inability or unwillingness to continue rehabilitation protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Generally recruited through the University of Utah Orthopaedic Center.
Groups:
- Standard of Care Intradiscal PRP Injections: There was only one group. All participants had standard-of-care intradiscal PRP injections.
Period: Overall Study
Arm/Group | Standard of Care Intradiscal PRP Injections
Started | 3
Completed | 0
Not Completed | 3
Not completed — The study was discontinued due to low enrollment. | 3

BASELINE CHARACTERISTICS:
Population: Baseline information was collected from 3 participants before the study was discontinued early.
Groups:
- Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections: There was only 1 group comprised of the 3 participants enrolled in the study before termination. All participants had standard-of-care intradiscal PRP injections.
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3
Height [Median (Full Range); unit: centimeters] | 185.4 [167.6 to 190.5]
Weight [Median (Full Range); unit: kilograms] | 87.5 [81.7 to 89.8]
Duration of Pain [Count of Participants; unit: Participants]
  1-2 years | 1
  3-5 years | 2
Radiologic Diagnosis Based on MRI of the Lumbar Spine? [Count of Participants; unit: Participants]
  Yes | 2
  No | 1
Numeric Rating Scale Low Back Pain Score [Median (Full Range); unit: units on a scale] — The Numeric Rating Scale was used to quantify low back pain by asking patients to rate their pain intensity on an 11-point scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
  units on a scale
    Current low back pain score | 4.0 [3.0 to 5.0]
    7-day average low back pain score | 3.0 [3.0 to 5.0]
Numeric Rating Scale Leg Pain Score [Median (Full Range); unit: units on a scale] — The Numeric Rating Scale (NRS) was used to quantify leg pain at baseline by asking patients to rate their pain intensity on an 11-point scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable".
  units on a scale
    Current leg pain score | 1.0 [0.0 to 3.0]
    7-day average leg pain score | 2.0 [0.0 to 2.0]
Oswestry Disability Index Score [Median (Full Range); unit: units on a scale] — The Oswestry Disability Index (ODI) is an instrument used in clinical and research applications to quantify disability due to low back pain as a percentage score (0-100%) based on patients' self-reported level of function in activities of daily living, with higher scores indicating greater disability.
  units on a scale | 9.0 [8.0 to 17.0]
Pain and Sleep Questionnaire 3-Item Index (PSQ-3) Score [Median (Full Range); unit: units on a scale] — The 3-Item Pain and Sleep Questionnaire is an instrument used in clinical and research applications to measure the impact of pain on sleep in chronic pain populations. A higher total score (range 0 to 300) indicates a greater extent of pain-related sleep interference.
  units on a scale | 190.0 [21.0 to 237.0]
PROMIS PF CAT Score [Median (Full Range); unit: units on a scale] — Patient-Reported Outcomes Measurement Information System Physical Function Computerized Adaptive Testing (PROMIS PF CAT) measures limitations of physical activity on a scale of 0 to 100, with higher scores indicating fewer limitations.
  units on a scale | 42.3 [35.5 to 50.4]
PROMIS Global Health Score [Median (Full Range); unit: units on a scale] — Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health is an instrument used in clinical and research applications to provide a general assessment of health across a variety of domains. Higher scores (range 0 to 100) indicate better overall health status.
  units on a scale | 33.0 [28.0 to 45.0]
Medication Quantification Scale (MQS) III Score [Median (Full Range); unit: units on a scale] — The Medication Quantification Scale (MQS) III is used to objectively quantify and monitor pain medication use (including opioid and non-opioid medications) in chronic pain populations. The lowest possible MQS III score is 0, indicating no current usage of any analgesic drugs assessed by this instrument. It is not possible to define a maximum score value because no theoretical upper limit exists. However, higher scores reflect greater negative impacts of a pain medication regimen, and a score of 6.8 points on the MQS III is comparable to 10 daily morphine equivalents in milligrams.
  units on a scale | 10.2 [0 to 21.4]
Daily Morphine Equivalent Dose [Median (Full Range); unit: milligrams of morphine] — Daily Morphine Equivalent Dose represents the amount of opioid medications that a patient is currently taking for pain, expressed as a common unit (milligrams of morphine).
  milligrams of morphine | 0.0 [0.0 to 0.0]

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale for Low Back Pain at 2-Month Follow-up
Description: Proportion of participants with ≥80% and ≥50% reductions from baseline in 7-day average low back pain intensity scores on the Numeric Rating Scale (NRS) at the 2-month follow-up assessment.
Time Frame: 2 months
Population: Presented here are primary outcome data collected from the 3 participants before the study was discontinued due to very low enrollment numbers.
Measure: Count of Participants; unit: Participants
Groups:
- Standard-of-care Intradiscal PRP Injections: There was only 1 group. All participants had standard-of-care intradiscal PRP injections
Arm/Group | Standard-of-care Intradiscal PRP Injections
Number analyzed (Participants) | 3
Participants
  Proportion of participants with ≥80% reduction in low back pain NRS score | 2
  Proportion of participants with ≥50% reduction in low back pain NRS score | 2

2. Secondary Outcome: Median Change in Low Back Pain Numeric Rating Scale (NRS) Score
Description: The Numeric Rating Scale (NRS) was used to quantify low back pain by asking patients to rate their pain intensity on an 11-point scale ranging from 0 to 10, with 0 representing "no pain at all" and 10 representing "the worst pain imaginable". NRS change scores were calculated by subtracting baseline scores from follow-up scores, so that negative change scores correspond to decreases in low back pain.
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: One participant did not complete the 1-month assessment and was lost to follow-up after the 2-month assessment. For the remaining 2 participants, outcome data were collected at all follow-up time points through 2 years before the study was discontinued for low enrollment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Standard of Care Intradiscal PRP Injections
Number analyzed (Participants) | 3
units on a scale
  1 month: number analyzed (Participants) | 2
  1 month | -1 [-1 to -1]
  2 months | -3 [-4 to -1]
  3 months: number analyzed (Participants) | 2
  3 months | -2 [-3 to -1]
  6 months: number analyzed (Participants) | 2
  6 months | -2 [-3 to -1]
  9 months: number analyzed (Participants) | 2
  9 months | -2 [-2 to -2]
  12 months: number analyzed (Participants) | 2
  12 months | -3 [-3 to -3]
  24 months: number analyzed (Participants) | 2
  24 months | -3 [-3 to -3]
  36 months: number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Patients With ≥30% Improvement From Baseline on the Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) is an instrument used in clinical and research applications to quantify disability due to low back pain as a percentage score based on patients' self-reported level of function in activities of daily living.
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: No ODI scores were recorded at the 1-month assessment. One participant was lost to follow-up after the 2-month assessment. For the remaining 2 participants, outcome data were collected at all follow-up time points through 2 years before the study was discontinued for low enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
Participants
  1 month: number analyzed (Participants) | 0
  2 months | 2
  3 months: number analyzed (Participants) | 2
  3 months | 1
  6 months: number analyzed (Participants) | 2
  6 months | 1
  9 months: number analyzed (Participants) | 2
  9 months | 2
  12 months: number analyzed (Participants) | 2
  12 months | 2
  24 months: number analyzed (Participants) | 2
  24 months | 2
  36 months: number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients With a ≥6 Score on Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change is a scale which measures participant reported satisfaction after an intervention. The outcome was measured as the percent of patients reporting a PGIC score of 6-7 (indicating "much improved" and "very much improved").
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
Participants
  1 month: number analyzed (Participants) | 2
  1 month | 1
  2 months | 2
  3 months: number analyzed (Participants) | 2
  3 months | 1
  6 months: number analyzed (Participants) | 2
  6 months | 2
  9 months: number analyzed (Participants) | 2
  9 months | 2
  12 months: number analyzed (Participants) | 2
  12 months | 2
  24 months: number analyzed (Participants) | 2
  24 months | 2
  36 months: number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Patients With a Medication Quantification Scale (MQS) III Score Reduction From Baseline of ≥6.8 Points
Description: A score of 6.8 points on the MQS III is equivalent to approximately 10 daily morphine equivalents
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
Participants
  1 month: number analyzed (Participants) | 2
  1 month | 2
  2 months | 1
  3 months: number analyzed (Participants) | 2
  3 months | 2
  6 months: number analyzed (Participants) | 2
  6 months | 2
  9 months: number analyzed (Participants) | 2
  9 months | 2
  12 months: number analyzed (Participants) | 2
  12 months | 2
  24 months: number analyzed (Participants) | 2
  24 months | 2
  36 months: number analyzed (Participants) | 0

6. Secondary Outcome: Oswestry Disability Index (ODI) Change Scores
Description: The Oswestry Disability Index (ODI) is an instrument used in clinical and research applications to quantify disability due to low back pain as a percentage score (0-100%) based on patients' self-reported level of function in activities of daily living, with higher scores indicating greater disability. ODI change scores were calculated by subtracting baseline scores from follow-up scores, so that negative change scores correspond to functional improvements.
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 3
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
score on a scale
  1 month: number analyzed (Participants) | 0
  2 months | -9.0 [-12.0 to 2.0]
  3 months: number analyzed (Participants) | 2
  3 months | -4.0 [-12.0 to 4.0]
  6 months: number analyzed (Participants) | 2
  6 months | -6.5 [-13.0 to 0.0]
  9 months: number analyzed (Participants) | 2
  9 months | -8.0 [-12.0 to -4.0]
  12 months: number analyzed (Participants) | 2
  12 months | -9.5 [-13.0 to -6.0]
  24 months: number analyzed (Participants) | 2
  24 months | -9.5 [-11.0 to -8.0]
  36 months: number analyzed (Participants) | 0

7. Secondary Outcome: PROMIS PF CAT Change Scores
Description: Patient-Reported Outcomes Measurement Information System Physical Function Computerized Adaptive Testing (PROMIS PF CAT) measures limitations of physical activity on a scale of 0 to 100, with higher scores indicating fewer limitations. PROMIS PF CAT change scores were calculated by subtracting baseline scores from follow-up scores, so that positive change scores represent improvements to functional limitations.
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
score on a scale
  1 month: number analyzed (Participants) | 2
  1 month | 6.3 [5.1 to 7.4]
  2 months | 12.5 [-1.6 to 25.2]
  3 months: number analyzed (Participants) | 2
  3 months | 6.2 [-0.1 to 12.5]
  6 months: number analyzed (Participants) | 2
  6 months | 11.3 [-2.4 to 24.9]
  9 months: number analyzed (Participants) | 2
  9 months | 8.7 [4.4 to 13.0]
  12 months: number analyzed (Participants) | 2
  12 months | 11.6 [9.1 to 14.1]
  24 months: number analyzed (Participants) | 2
  24 months | 15.9 [14.1 to 17.7]
  36 months: number analyzed (Participants) | 0

8. Secondary Outcome: Pain and Sleep Questionnaire 3-Item Index (PSQ-3) Change Scores
Description: The 3-Item Pain and Sleep Questionnaire is an instrument used in clinical and research applications to measure the impact of pain on sleep in chronic pain populations. A higher total score (range 0 to 300) indicates a greater extent of pain-related sleep interference. PSQ-3 change scores were calculated by subtracting baseline scores from follow-up scores, so that negative change scores correspond to reductions in pain-related sleep interference.
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
score on a scale
  1 month: number analyzed (Participants) | 2
  1 month | -175.0 [-220.0 to -130.0]
  2 months | -111.0 [-187.0 to -21.0]
  3 months: number analyzed (Participants) | 2
  3 months | -153.0 [-195.0 to -111.0]
  6 months: number analyzed (Participants) | 2
  6 months | -163.0 [-170.0 to -156.0]
  9 months: number analyzed (Participants) | 2
  9 months | -186.5 [-233.0 to -140.0]
  12 months: number analyzed (Participants) | 2
  12 months | -178.5 [-237.0 to -120.0]
  24 months: number analyzed (Participants) | 2
  24 months | -200.5 [-231.0 to -170.0]
  36 months: number analyzed (Participants) | 0

9. Secondary Outcome: Patient Satisfaction Scores
Description: The Patient Satisfaction Score represents patient satisfaction with the healthcare received using a five-point Likert scale where 1 = "very dissatisfied"; 2 = "dissatisfied"; 3 = "neither satisfied nor dissatisfied"; 4 = "satisfied"; and 5 = "very satisfied".
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
score on a scale
  1 month | 5.0 [5.0 to 5.0]
  2 months | 5.0 [4.0 to 5.0]
  3 months: number analyzed (Participants) | 2
  3 months | 4.5 [4.0 to 5.0]
  6 months: number analyzed (Participants) | 2
  6 months | 5.0 [5.0 to 5.0]
  9 months: number analyzed (Participants) | 2
  9 months | 5.0 [5.0 to 5.0]
  12 months: number analyzed (Participants) | 2
  12 months | 5.0 [5.0 to 5.0]
  24 months: number analyzed (Participants) | 2
  24 months | 5.0 [5.0 to 5.0]
  36 months: number analyzed (Participants) | 0

10. Secondary Outcome: Patient Global Impression of Change (PGIC) Scores
Description: Patient Global Impression of Change (PGIC) scores represent participants' overall satisfaction after an intervention. Participants are asked to rate their perception of change on a scale of 1 to 7, where 1="very much worse", 2="much worse", 3="worse", 4="no change", 5="improved", 6="much improved", and 7="very much improved".
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
score on a scale
  1 month: number analyzed (Participants) | 2
  1 month | 6.5 [6.0 to 7.0]
  2 months | 6.0 [5.0 to 7.0]
  3 months: number analyzed (Participants) | 2
  3 months | 6.0 [5.0 to 7.0]
  6 months: number analyzed (Participants) | 2
  6 months | 6.5 [6.0 to 7.0]
  9 months: number analyzed (Participants) | 2
  9 months | 7.0 [7.0 to 7.0]
  12 months: number analyzed (Participants) | 2
  12 months | 7.0 [7.0 to 7.0]
  24 months: number analyzed (Participants) | 2
  24 months | 7.0 [7.0 to 7.0]
  36 months: number analyzed (Participants) | 0

11. Secondary Outcome: Opioid Consumption in Daily Morphine Equivalents
Time Frame: 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 24 months, 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: milligrams of morphine
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
milligrams of morphine
  1 month: number analyzed (Participants) | 2
  1 month | 0 [0 to 0]
  2 months | 0 [0 to 0]
  3 months: number analyzed (Participants) | 2
  3 months | 0 [0 to 0]
  6 months: number analyzed (Participants) | 2
  6 months | 0 [0 to 0]
  9 months: number analyzed (Participants) | 2
  9 months | 0 [0 to 0]
  12 months: number analyzed (Participants) | 2
  12 months | 0 [0 to 0]
  24 months: number analyzed (Participants) | 2
  24 months | 0 [0 to 0]
  36 months: number analyzed (Participants) | 0

12. Secondary Outcome: Proportion of Patients Who Underwent Lumbar Spinal Surgery During the Study Period
Time Frame: 24 months, 36 months
Population: The study was discontinued for low enrollment prior to the 36-month endpoint. No study participants had undergone lumbar spinal surgeries as of the latest follow-up assessment (24 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Intradiscal Platelet-Rich Plasma (PRP) Injections
Number analyzed (Participants) | 3
Participants
  24 months | 0
  36 months: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 36 months
Description: The rate of SAE's or deaths from this procedure is very low. "Utilizing fluoroscopy, the risk of nerve damage, spinal cord injury or intravascular injection is less than 1:500,000" (protocol page 5)
Arm/Group | Standard-of-care Intradiscal PRP Injections
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The single greatest limitation is that the study was ended early due to extremely low participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT04544709/Prot_SAP_000.pdf